CLINICAL TRIAL: NCT06200311
Title: Atrial Fibrillation (AF) Ablation to Prevent Disease Progression of AF-induced Atrial Cardiomyopathy in Women and Men
Acronym: RACE X
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RACE X trial
Record Dates: First submitted 2023-12-01; First posted 2024-01-11 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Fibrillation, Atrial; Atrial Cardiomyopathy
Keywords: pulmonary vein isolation; mHealth; atrial fibrillation; atrial cardiomyopathy; AF ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Eligible patients with ACMP and AF will be randomised to AF ablation and pharmacological rhythm management
Who Masked: Outcomes Assessor
Masking Description: endpoints will be adjudicated by a blinded clinical endpoint committee
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AF ablation (Experimental): These patients will undergo Pulmonary vein isolation (PVI) (only)
  Interventions: Procedure: Pulmonary vein isolation
- Pharmacological rhythm management (Active Comparator): These patients will take rate control medication. If this therapy fails, pharmacological rhythm control and AF ablation are 2nd and 3rd line options respectively within this arm,
  Interventions: Drug: Pharmacological rhythm management

INTERVENTIONS:
Procedure: Pulmonary vein isolation — Pulmonary vein isolation using pulsed field ablation (PFA), cryoballoon or radiofrequency ablation (RFA)
  Other Names: AF ablation
  Arms: AF ablation
Drug: Pharmacological rhythm management — 1st line: rate control, 2nd line: pharmacological rhythm management. 3rd line: AF ablation
  Arms: Pharmacological rhythm management

SUMMARY:
The goal of clinical trial is to compare AF ablation to pharmacological rhythm management (being rate or rhythm control) in AF patients with signs of atrial cardiomyopathy (as defined by left atrial volume index >34 ml/m2) The main objective it aims to answer is to determine whether AF ablation compared to pharmacological rhythm management in ACMP patients with AF reduces the incidence of the composite primary endpoint of CV death and first CV hospitalization/urgent visit.

DETAILED DESCRIPTION:
The RACE X trial investigates the impact of atrial cardiomyopathy (ACMP) and ablation timing on adverse outcomes in atrial fibrillation (AF) patients. ACMP leads to an atrial substrate less responsive to rhythm control, exacerbating AF recurrence and progression. This trial assesses whether AF ablation versus pharmacological rhythm management reduces the combined primary endpoint of cardiovascular (CV) death and hospitalization in ACMP and AF patients. Secondary objectives include measuring ACMP progression, ACMP-related outcomes, mortality, hospitalizations, AF symptoms, quality of life, and healthcare costs. Exploratory goals involve various additional measurements. This prospective, multicenter, open-label, blinded-endpoint, phase IIIb trial randomizes patients with ACMP and AF to receive either AF ablation or pharmacological rhythm management. Follow-up involves mobile health (mHealth) applications, questionnaires, and heart rhythm monitoring across 13 Dutch hospitals. Ineligible patients undergoing AF ablation join an observational registry. The trial population consists of patients aged 65-80 years with confirmed ACMP and ECG-confirmed AF. With 604 patients and a median 2.5-year follow-up, the trial aims to assign patients equally to each intervention. The primary endpoint is a composite of CV death and hospitalization. Catheter ablation, a safe and efficient technique, minimizes patient burden, and remote follow-up through mHealth reduces site visits. Additional study procedures are integrated into routine care, ensuring a streamlined process.

ELIGIBILITY:
Inclusion criteria

* Confirmed ACMP (LAVI >34 ml/m2)
* ECG-confirmed AF
* Age: 65-80 years old
* Patients eligible for both treatment strategies judged by the treating physician signed and dated informed consent prior to admission to the trial

Exclusion criteria

* Longstanding (>1 year) persistent or permanent (accepted) AF
* Previous left atrial (LA) ablation or LA surgery
* AF due to a reversible cause (e.g. hyperthyroidism, post-operative AF)
* Recent (<90 days) acute coronary syndrome, stroke/TIA or cardiac intervention (Cardiac interventions include percutaneous coronary intervention, coronary artery bypass grafting, and heart valve repair or replacement (endovascular or surgical))
* Intracardiac thrombus
* HF NYHA III/IV
* Impaired renal function, defined as estimated glomerular filtration rate ≤25 ml/min/1.73m2
* Presence of (or scheduled for) mechanical assist device or heart transplant
* Severe aortic or mitral valve disease
* Complex congenital heart disease
* Life expectancy <1 year
* Currently enrolled in another clinical randomized trial

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — 1:1 by stratitification
Enrollment: 604 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2029-07-25 (Estimated); Study Completion 2029-07-25 (Estimated)

PRIMARY OUTCOMES:
A composite of cardiovascular (CV) death and first CV hospitalisation/urgent visit. | through study completion, a median of 2.5 years
  Atrial cardiomyopathy (ACMP)-associated complications

SECONDARY OUTCOMES:
ACMP progression or regression | through study completion, a median of 2.5 years
  As measured by LAVI (left atrial volume index) increase or decrease
Hospitalisations/urgent visits for AF, atrial flutter (AFL) or atrial tachycardia (AT) | through study completion, a median of 2.5 years
  Hospitalisations/urgent visits for AF, AFL or AT
Hospitalisations/urgent visits for heart failure (HF) | through study completion, a median of 2.5 years
  Hospitalisations/urgent visits for heart failure
Hospitalisations/urgent visits for ischemic stroke (including transient ischemic attack (TIA)) | through study completion, a median of 2.5 years
  Hospitalisations/urgent visits for ischemic stroke (including TIA)
Cardiovascular death | through study completion, a median of 2.5 years
  Cardiovascular death
All-cause mortality | through study completion, a median of 2.5 years
  All-cause mortality
Symptoms and improve quality of life (QoL) measured by EuroQol-5D-5L questionnaire. (higher score indicating a better QoL) | through study completion, a median of 2.5 years
Symptoms and improve quality of life (QoL) measured by Atrial Fibrillation Effect on Quality of Life (AFEQT) questionnaire (higher score indicating less symptoms and a better QoL) | through study completion, a median of 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Michiel Rienstra, Prof. dr., Principal Investigator — University Medical Center Groningen
Locations (1):
- UMCG, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No